CLINICAL TRIAL: NCT05194449
Title: Nonpharmacologic Reduction of Periprocedural Pain, Anxiety, and Prescription Drug Use Phase II
Brief Title: Nonpharmacologic Reduction of Periprocedural Pain and Anxiety in Dentistry
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started since the study was not funded
Sponsor: Hypnalgesics, LLC (Industry)
Collaborators: Cambridge Health Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: R44AT009517
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Dental Anxiety; Dental Pain; Root Work
Keywords: Nonpharmacologic analgesia; Medical app; Relaxation; Hypnosis
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Intervention Model Description: This is a single-blind placebo-controlled trial comparing a Comfort Talk® calmative app (Cft Group) with a white noise app (WN, Control Group).
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Two iPad tablets used in the study will be labeled A and B and will be preloaded with the app or white noise by the Hypnalgesics, LLC in randomized sequence. Personnel at CHA will not be aware which tablet presents test or control content. The opening screen and option screen of the white noise control app will use the same color scheme and lay-out as the one of the test Comfort Talk app. The statistical team will receive the encoded data entries and will not be informed about the content of the tablets until all analyses are completed. Since they also will not have direct contact with the study patients they are also not at risk of becoming unblinded during app use by the patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comfort Talk® App (Cft) Group (Experimental): Mobile app with elements of relaxation, self-hypnosis, and reframing of distress
  Interventions: Other: Comfort Talk® App
- Placebo Group (Placebo Comparator): Mobile app with white noise choices having the same looks and functionality as the active Comfort Talk® 1st app
  Interventions: Other: Placebo App

INTERVENTIONS:
Other: Comfort Talk® App — Patients will receive a tablet preloaded with the Comfort Talk® app in the dental waiting room on an intent-to-treat basis. They can listen as much or as little as they wish during waiting and during their dental treatment. Upon departure, they will receive a download coupon for the app for home use.
  Other Names: Self-hypnotic relaxation app; Test app
  Arms: Comfort Talk® App (Cft) Group
Other: Placebo App — Patients will receive a tablet preloaded with a white noise app in the dental waiting room on an intent-to-treat basis. They can listen as much or as little as they wish during waiting and during their dental treatment.
  Other Names: White noise app
  Arms: Placebo Group

SUMMARY:
Dental pain and anxiety are usually managed by local anesthetics and sedatives, but patient anxiety and fear of pain remain common and adversely affect oral health behavior and outcomes. The long-term goal is to provide a validated behavioral alternative/adjunct for managing dental anxiety and pain through a commercial Comfort Talk® (Cft) app. Such an application should benefit the patients undergoing the >300 million dental procedures per year in the US alone. In Phase I (Clinical Trials Identifier NCT03328208), the investigators designed such an app based on short Comfort Talk® scripts and snippets that, when spoken live by trained personnel in our prior large-scale clinical trials, reduced pain, anxiety, and drug use during invasive procedures, and when used practice-wide, improved patient attendance, throughput, and economics. In Phase I, the Cft app significantly reduced pain and anxiety in the dental waiting room. In Phase II, the investigators propose to further assess its impact.

We hypothesize that:

* The Cft app reduces pain and anxiety in the waiting room
* The Cft app improves the patient experience and cooperation during dental treatment
* The Cft app improves operations and economics of dental practices
* Heart rate tracings are helpful in identifying outcome-critical app elements

  150 patients scheduled for root canals or dental implants will receive in randomized sequence the Cft app or a placebo white noise app in the dentistry waiting room of Cambridge Health Alliance. Anxiety and pain will be measured subjectively on validated scales (0-no anxiety/no pain at all; 10-worst anxiety/pain possible) before listening and throughout the visit. Heart rate (HR) and ECG will be continuously recorded to assess adverse events and, in the absence of a validated biomarker for pain and anxiety, serve as an exploratory physiologic indicator of distress. Usage patterns of the Cft and the placebo apps will be established electronically through time-stamped background capture, de-identified, and uploaded to a database along with the corresponding HR recordings and overlayed with the patient's subjective ratings and procedure steps to identify outcome-critical elements of the app.

We will record chair-time, staff-time, use of anesthetics and sedatives, if applicable, and patient and staff satisfaction, supplemented by bulk data acquired from other practices that use a co-branded version of the app, to determine the economic impact of the Cft app.

DETAILED DESCRIPTION:
Dental pain and anxiety are usually managed by local anesthetics and sedatives, but patient anxiety and fear of pain remain common and adversely affect oral health behavior and outcomes. The long-term goal is to provide a validated behavioral alternative/adjunct for managing dental anxiety and pain through a commercial Comfort Talk® (Cft) app. Such an application should benefit the patients undergoing the >300 million dental procedures per year in the US alone. In Phase I (Clinical Trials Identifier NCT03328208), the investigators designed such an app based on short Comfort Talk® scripts and snippets that, when spoken live by trained personnel in their prior large-scale clinical trials, reduced pain, anxiety, and drug use during invasive procedures, and when used practice-wide, improved patient attendance, throughput, and economics. In Phase I, the Cft app significantly reduced pain and anxiety in the dental waiting room. In Phase II, the investigators propose to further assess its impact. In Phase II, the investigators propose to further assess the impact of the Cft app in dentistry in accordance with an objective of the National Center for Complementary and Integrative Health(NCCIH) 2021-2025 Strategic Plan: testing the integration of a complementary approach into healthcare in a real-world setting.

The hypotheses are:

* The Cft app reduces pain and anxiety in the waiting room
* The Cft app improves the patient experience and cooperation during dental treatment
* The Cft app improves operations and economics of dental practices
* Heart rate tracings are helpful in identifying outcome-critical app elements

  150 patients scheduled for root canals or dental implants will receive in randomized sequence the Cft app or a placebo white noise app in the dentistry waiting room.

The trial will be performed at Cambridge Health Alliance (CHA), Department of Dental Medicine, based on their high patient volume (>12,000 annual visits) and ethnically/racially diverse mix of patients. CHA is a nationally respected and innovative healthcare system and Massachusetts' largest safety net organization. CHA is committed to providing care for the undeserved and promoting interprofessional/cross-disciplinary care for all regardless of cultural, racial, or socioeconomic background. All patients of the dental clinic also receive their primary care through CHA, enabling electronic chart review regarding prior dental experiences, vital signs, and medical history.

The study will be carried out in accordance with an intent-to-treat comparison of the effects of a self-hypnotic relaxation Comfort Talk® (Cft) app versus a White Noise (WN), placebo-control app delivered through tablet in the dental waiting room. The comparison of test versus placebo apps is rare in the literature and enhances the rigor of the study. The same look and functionality of the Cft and WN apps will allow for as much blinding of the staff as physically feasible. The tablets' covers have A and B stickers with the designation for Cft and WN randomly determined. A research assistant (RA) will ask eligible patients to participate, consent, and fill out the patient's history based on the electronic record and patients' verbal information, and obtain their levels of pain and anxiety on a timed intake sheet. While patients fill out an anxiety questionnaire the RA retrieves and opens a sealed randomization envelope. The RA helps the patient to place an upper sternal patch for placement of a small ECG/heart rate monitor, hands them the assigned tablet, and goes over a print-out visual of generic tablet instructions to assure patients understand the usage of the apps without having to open the tablet to reveal their nature. The RA then invites the patient to engage with the assigned application as they like during the entire duration of their visit.

The RA keeps track of the time and the following data: pain and anxiety at baseline, at the end of the waiting room time, after entry in the treatment room, then every 10 minutes of the treatment, and at the end of the procedure; start of the treatment and steps such as use of a drill, anesthetics, or sedation if applicable, adverse events, and number and type of dental staff present. Upon treatment completion, patients and staff will fill out satisfaction with treatment questionnaires.

In the background, de-identified usage patterns of the Cft and WN apps will be electronically recorded through time-stamped capture. For analysis, they will be overlayed with the patient's timed subjective ratings and the electronically obtained heart rate data to identify outcome-critical elements of the app. This data will help identify the most beneficial app features which will provide the investigators with a unique opportunity to describe and better understand non-pharmacological interventions in general and will help inform future studies.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo a root canal or dental implant procedure at Cambridge - Health Alliance
* Able to hear, write and read in English, as the ComfortTalk® scripts, study scales and take-home diary are in English
* Able to operate a standard smart tablet
* Willing and able to give informed consent

Exclusion Criteria:

* Known acute psychiatric disorder, such as multiple personalities which will be assessed on the medical history form
* Implanted cardiac medical device
* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety during the dental visit (Change as Compared to Beginning of the Waiting Room Time) | Up to 180 minutes
  Anxiety as measured by self-report on a 0-10 scale with 0=no anxiety at all and 10=worst anxiety possible; change from the beginning to the end of the waiting room time, measured before listening to the app, at the end of the waiting room, every 10 minutes on the dental chair, and after treatment completion
Pain during the dental visit (Change as Compared to Beginning of the Waiting Room Time) | Up to 180 minutes
  Pain as measured by self-report on a 0-10 scale with 0=no pain at all and 10=worst pain possible; change from the beginning to the end of the waiting room time, measured before listening to the app, at the end of the waiting room, every 10 minutes on the dental chair, and after treatment completion

SECONDARY OUTCOMES:
Adverse events | Up to 180 minutes
  Observable adverse events such as fainting, hemodynamics instability and those detected post visit by analysis of ECG/heart rate recordings (de novo bradycardia, tachycardia, arrhythmia, abnormal ECG changes)
Chair Time | Up to 180 minutes
  The time the patient will be on the dental treatment chair
Staff Time | Up to 180 minutes
  How long and which kind of staff personnel interacted with the patient during the visit (e.g., dentist, assistant, secretary) for assessment of the economic impact.
Patient Satisfaction | 10 minutes
  The survey uses a 1-5 scale (1=very poor, 5=very well) and asks how the staff treated the patient, how well the staff worked together to provide care, how well the patient's pain was controlled, how well the staff did everything to help with their pain, how to rate the overall care, how well the tablet affected the way the patient felt, and whether the patient would recommend the facility.
Staff Satisfaction | 10 minutes
  Staff assessment will use a questionnaire piloted in Phase I assessing technical difficulty of the dental treatment, patient cooperation, perceived patient comfort, staff comfort, help perceived by app use, and overall staff satisfaction on a 1-4 Likert scale (not at all, a little, somewhat, a lot).

CONTACTS AND LOCATIONS:
Overall Officials: Evira V Lang, MD, Principal Investigator — Hypnalgesics, LLC d/b/a Comfort Talk®

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang EV, Jackson W, Senn P, Aroni DKK, Finkelman MD, Corino TA, Conway G, Kulich RJ. Efficacy of a Self-Hypnotic Relaxation App on Pain and Anxiety in a Randomized Clinical Trial: Results and Considerations on the Design of Active and Control Apps. Int J Clin Exp Hypn. 2021 Apr-Jun;69(2):277-295. doi: 10.1080/00207144.2021.1883988. Epub 2021 Mar 16. PMID 33724898
- [Background] Lang EV, Benotsch EG, Fick LJ, Lutgendorf S, Berbaum ML, Berbaum KS, Logan H, Spiegel D. Adjunctive non-pharmacological analgesia for invasive medical procedures: a randomised trial. Lancet. 2000 Apr 29;355(9214):1486-90. doi: 10.1016/S0140-6736(00)02162-0. PMID 10801169
- [Background] Lang EV, Berbaum KS, Faintuch S, Hatsiopoulou O, Halsey N, Li X, Berbaum ML, Laser E, Baum J. Adjunctive self-hypnotic relaxation for outpatient medical procedures: a prospective randomized trial with women undergoing large core breast biopsy. Pain. 2006 Dec 15;126(1-3):155-64. doi: 10.1016/j.pain.2006.06.035. Epub 2006 Sep 7. PMID 16959427
- [Background] Lang EV, Berbaum KS, Pauker SG, Faintuch S, Salazar GM, Lutgendorf S, Laser E, Logan H, Spiegel D. Beneficial effects of hypnosis and adverse effects of empathic attention during percutaneous tumor treatment: when being nice does not suffice. J Vasc Interv Radiol. 2008 Jun;19(6):897-905. doi: 10.1016/j.jvir.2008.01.027. Epub 2008 Mar 17. PMID 18503905
- [Background] Lang EV, Tan G, Amihai I, Jensen MP. Analyzing acute procedural pain in clinical trials. Pain. 2014 Jul;155(7):1365-1373. doi: 10.1016/j.pain.2014.04.013. Epub 2014 Apr 13. PMID 24731852